CLINICAL TRIAL: NCT04066842
Title: Evaluation Of Vitamin D In Systemic Sclerosis Patients With Periodontitis: A Possible Role In Cardiovascular Disease Risk Progression?
Brief Title: Vitamin D in Systemic Sclerosis Patients With Periodontitis
Status: Completed | Type: Observational
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Gaetano Isola, DDS, PhD, Junior Assistant Professor, University of Messina
Other Study IDs: 10-918
Record Dates: First submitted 2019-08-22; First posted 2019-08-26 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1 - Controls: Control Healthy controls
  Interventions: Other: Observation
- 2 - SSc: SSc Systemic Sclerosis
  Interventions: Other: Observation
- 3 - Cardiovascular: Cardiovascular Cardiovascular disease
  Interventions: Other: Observation
- 4 - SSc+Periodontitis: SSc+ Periodontitis Systemic Sclerosis with Periodontitis
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Evaluation of Vitamin D levels and correlation of Vitamin D levels level with periodontal and cardiovascular disease

SUMMARY:
Vitamin D has been considered to possess anti-inflammatory and antimicrobial activity which may be a link for the known interaction of Systemic Sclerosis (SSc) and coronary heart disease (CHD). This study investigated the association between serum vitamin D levels and SSc and periodontitis in patients with SSc, CP and with CHD.

Furthermore, the objective was to determine if periodontitis and CHD had an impact on serum vitamin D levels.

DETAILED DESCRIPTION:
Using a cross-sectional design, a total of 42 patients with SSc, 43 patients with CHD, 41 patients with both SSc and CP, and 42 healthy patients were enrolled in the present study.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least twenty teeth
* CP with a minimum of 40% of sites with a clinical attachment level (CAL)

  ≥2mm and probing depth (PD) ≥4mm;
* Presence of at least ≥2 mm of crestal alveolar bone loss verified on digital periapical radiographs
* Presence of ≥40% sites with bleeding on probing (BOP)

Exclusion Criteria:

* Intake of contraceptives
* Intake of immunosuppressive or anti-inflammatory drugs throughout the last three months prior to the study
* Status of pregnancy or lactation
* Previous history of excessive drinking
* Allergy to local anaesthetic
* Intake of drugs that may potentially determine gingival hyperplasia such as Hydantoin, Nifedipine, Cyclosporin A or similar drugs.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 42 patients with SSc, 43 patients with CHD, 41 patients with both SSc and CP, and 42 healthy patients were enrolled in the present study
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Vitamin D levels | 1 year
  Evaluation of serum Vitamin D levels

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — University of Catania
Locations (1):
- University of Messina, Messina, Italy

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Public register
Access Criteria: Policlinic Messina website